CLINICAL TRIAL: NCT02296541
Title: A Phase 1 Randomized, Double-Blind, Placebo Controlled Clinical Trial to Evaluate the Safety and Immunogenicity of 3 Different HIV-1 DNA Priming Regimens (Nat-B Env, CON-S Env, and Mosaic Env) With MVA-CMDR Boosts in Healthy, HIV-1-Uninfected Adults
Brief Title: Evaluating the Safety and Immune Response to Three Different DNA HIV Vaccines Administered With a MVA-CMDR Boost Vaccine in Healthy, HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: CHAVI (Unknown); IPPOX Foundation (Other); MHRP (Unknown); HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 106; 11999 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1: DNA Nat-B env and MVA-CMDR (Experimental): Participants will receive a single injection of DNA Nat-B env at Months 0, 1, and 2. They will receive a single injection of MVA-CMDR at Months 4 and 8.
  Interventions: Biological: DNA Nat-B env; Biological: MVA-CMDR
- Group 1: Placebo vaccines for DNA Nat-B env and MVA-CMDR (Placebo Comparator): Participants will receive a single injection of placebo for DNA Nat-B env at Months 0, 1, and 2. They will receive a single injection of placebo for MVA-CMDR at Months 4 and 8.
  Interventions: Biological: Placebo for DNA Nat-B env; Biological: Placebo for MVA-CMDR
- Group 2: DNA CON-S env and MVA-CMDR (Experimental): Participants will receive a single injection of DNA CON-S env at Months 0, 1, and 2. They will receive a single injection of MVA-CMDR at Months 4 and 8.
  Interventions: Biological: DNA CON-S env; Biological: MVA-CMDR
- Group 2: Placebo vaccines for DNA CON-S env and MVA-CMDR (Placebo Comparator): Participants will receive a single injection of placebo for DNA CON-S env at Months 0, 1, and 2. They will receive a single injection of placebo for MVA-CMDR at Months 4 and 8.
  Interventions: Biological: Placebo for DNA CON-S env; Biological: Placebo for MVA-CMDR
- Group 3: DNA Mosaic env and MVA-CMDR (Experimental): Participants will receive a single injection of DNA Mosaic env at Months 0, 1, and 2. They will receive a single injection of MVA-CMDR at Months 4 and 8.
  Interventions: Biological: DNA Mosaic env; Biological: MVA-CMDR
- Group 3: Placebo vaccines for DNA Mosaic env and MVA-CMDR (Placebo Comparator): Participants will receive a single injection of placebo for DNA Mosaic env at Months 0, 1, and 2. They will receive a single injection of placebo for MVA-CMDR at Months 4 and 8.
  Interventions: Biological: Placebo for DNA Mosaic env; Biological: Placebo for MVA-CMDR

INTERVENTIONS:
Biological: DNA Nat-B env — 4 mg to be administered as 1 mL intramuscularly (IM) by Biojector 2000® or with a needle and syringe in the deltoid muscle of the non-dominant arm (unless medically contraindicated)
  Arms: Group 1: DNA Nat-B env and MVA-CMDR
Biological: DNA CON-S env — 4 mg to be administered as 1 mL IM by Biojector 2000® or with a needle and syringe in the deltoid muscle of the non-dominant arm (unless medically contraindicated)
  Arms: Group 2: DNA CON-S env and MVA-CMDR
Biological: DNA Mosaic env — 4 mg to be administered as 1 mL IM by Biojector 2000® or with a needle and syringe in the deltoid muscle of the non-dominant arm (unless medically contraindicated)
  Arms: Group 3: DNA Mosaic env and MVA-CMDR
Biological: MVA-CMDR — 1×10^8 plaque forming units (pfu) to be administered as 1 mL IM in the deltoid muscle of the non-dominant arm (unless medically contraindicated)
  Other Names: Modified Vaccinia Virus Ankara (MVA-CMDR)
  Arms: Group 1: DNA Nat-B env and MVA-CMDR; Group 2: DNA CON-S env and MVA-CMDR; Group 3: DNA Mosaic env and MVA-CMDR
Biological: Placebo for DNA Nat-B env — Sodium Chloride for Injection, 0.9% to be administered as 1 mL IM by Biojector 2000® or with a needle and syringe in the deltoid muscle of the non-dominant arm (unless medically contraindicated)
  Arms: Group 1: Placebo vaccines for DNA Nat-B env and MVA-CMDR
Biological: Placebo for DNA CON-S env — Sodium Chloride for Injection, 0.9% to be administered as 1 mL IM by Biojector 2000® or with a needle and syringe in the deltoid muscle of the non-dominant arm (unless medically contraindicated)
  Arms: Group 2: Placebo vaccines for DNA CON-S env and MVA-CMDR
Biological: Placebo for DNA Mosaic env — Sodium Chloride for Injection, 0.9% to be administered as 1 mL IM by Biojector 2000® or with a needle and syringe in the deltoid muscle of the non-dominant arm (unless medically contraindicated)
  Arms: Group 3: Placebo vaccines for DNA Mosaic env and MVA-CMDR
Biological: Placebo for MVA-CMDR — Sodium Chloride for Injection, 0.9% to be administered as 1 mL IM in the deltoid muscle of the non-dominant arm (unless medically contraindicated)
  Arms: Group 1: Placebo vaccines for DNA Nat-B env and MVA-CMDR; Group 2: Placebo vaccines for DNA CON-S env and MVA-CMDR; Group 3: Placebo vaccines for DNA Mosaic env and MVA-CMDR

SUMMARY:
The purpose of this study is to evaluate the safety and immune response to three DNA vaccines and a MVA-CMDR vaccine that may boost the immune response to the DNA vaccines in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and immunogenicity to four different HIV vaccines in healthy, HIV-uninfected adults. The vaccines include three DNA vaccines-DNA Nat-B env, DNA CON-S env, and DNA Mosaic env-and a vaccine called MVA-CMDR that may boost the immune response to the DNA vaccines.

The study will enroll healthy, HIV-uninfected participants aged 18 to 50 years. Participants will be randomly assigned to one of three groups and will receive either one of the experimental vaccine regimens or a placebo vaccine regimen. Group 1 participants will receive the DNA Nat-B env and MVA-CMDR vaccines or placebo. Group 2 participants will receive the DNA CON-S env and MVA-CMDR vaccines or placebo. Group 3 participants will receive DNA Mosaic env and MVA-CMDR vaccines or placebo.

All participants will receive one of their assigned vaccines at study entry (Month 0), and Months 1, 2, 4, and 8.

Total study duration will be either 3 years after enrollment (for participants in the United States) or 5 years after enrollment (for participants in Switzerland). For all participants, study visits will occur at study entry (Month 0), and Months 0.5, 1, 1.5, 2, 2.5, 4, 4.5, 8, 8.25, 8.5, 11, 13.75, and 14. After the last study visit, participants will be contacted annually by phone or e-mail for a total of 3 (U.S. participants) or 5 (Switzerland participants) years to answer questions about their health.

All study visits will include a physical exam, HIV risk reduction counseling, and an interview and/or questionnaire. Select study visits will include blood collection, urine and stool collection, HIV testing, an electrocardiogram (ECG), and a pregnancy test for participants who were born female. For participants receiving the MVA-CMDR vaccine, select study visits may also include an assessment of cardiac symptoms.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: participant demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to be contacted annually after completion of scheduled clinic visits for a total of 3 years for U.S. participants (5 years for participants in Switzerland) following initial study injection
* Agrees not to enroll in another study of an investigational research agent
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit

Laboratory Inclusion Values

Hemogram/Complete Blood Count (CBC)

* Hemoglobin greater than or equal to 12.5 g/dL for participants who were born female, greater than or equal to 13.5 g/dL for participants who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry

* Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to the institutional upper limit of normal
* Cardiac Troponin T or I (cTnT or cTnI) does not exceed the institutional upper limit of normal

Virology

* Negative HIV-1 and -2 blood test: U.S. participants must have a negative Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA). Non-U.S. site may use locally available assays that have been approved by HVTN Laboratory Operations.
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range)

Reproductive Status

* Participants who were born female: negative serum or urine beta human chorionic gonadotropin (beta-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: participants who were born female must:

  * Agree to consistently use effective contraception (information on effective contraception methods can be found in the protocol) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit;
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.
* Participants who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit.

Exclusion Criteria:

General

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40
* Intent to participate in another study of an investigational research agent during the planned duration of the HVTN 106 study
* Pregnant or breastfeeding

Vaccines and Other Injections

* Smallpox vaccine received within the last 5 years
* HIV vaccine(s) received in a prior HIV vaccine trial. For participants who have received control/placebo in an HIV vaccine trial, the HVTN 106 Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis and the identity of the study control/placebo must be obtained.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For participants who have received control/placebo in an experimental vaccine trial, the HVTN 106 PSRT will determine eligibility on a case-by-case basis. For participants who have received an experimental vaccine(s) more than 5 years ago, eligibility for enrollment will be determined by the HVTN 106 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (e.g., tetanus, pneumococcal, hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

Immune System

* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses less than 2 mg/kg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment
* Serious adverse reactions to vaccines or to vaccine components such as neomycin or streptomycin, including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease
* Immunodeficiency
* Hypersensitivity to eggs and/or egg products

Clinically Significant Medical Conditions

* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion can be found in the protocol.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma exclusion criteria: Asthma other than mild, well-controlled asthma. More information on this criterion can be found in the protocol.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone (Not excluded: history of isolated gestational diabetes)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these participants, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up)
* Participants who have 2 or more of the following cardiac risk factors:

  * Participant report of history of elevated blood cholesterol defined as fasting low-density lipoprotein (LDL) greater than 160 mg/dL;
  * First degree relative (e.g., mother, father, brother, or sister) who had coronary artery disease before the age of 50 years;
  * Current smoker; or
  * BMI greater than or equal to 35
* Electrocardiogram (ECG) with clinically significant findings, or features that would interfere with the assessment of myo/pericarditis, as determined by the contract ECG Lab, cardiologist, or study clinician. More information on this criterion can be found in the protocol.
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded: participant who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past 3 years. Also exclude if participant has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2014-12; Primary Completion 2016-11 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Frequency of local and systemic injection site reactogenicity signs and symptoms for each type of vaccine | Measured through Month 8
Severity of local and systemic injection site reactogenicity signs and symptoms for each type of vaccine | Measured through Month 8
Frequency of adverse events (AEs) | Measured through participant follow-up (3 and 5 years for participants in the United States and Switzerland, respectively)
  Categorized by MedDRA body system, MedDRA preferred term, severity, and assessed relationship to study products; detailed description of all AEs meeting Division of AIDS (DAIDS) criteria for expedited reporting (EAE)
Laboratory measure of safety: measurement of white blood cells (WBC) | Measured through Month 8
Laboratory measure of safety: measurement of neutrophils | Measured through Month 8
Laboratory measure of safety: measurement of lymphocytes | Measured through Month 8
Laboratory measure of safety: measurement of hemoglobin | Measured through Month 8
Laboratory measure of safety: measurement of platelets | Measured through Month 8
Laboratory measure of safety: measurement of alanine aminotransferase (ALT) | Measured through Month 8
Laboratory measure of safety: measurement of aspartate aminotransferase (AST) | Measured through Month 8
Laboratory measure of safety: measurement of alkaline phosphatase | Measured through Month 8
Laboratory measure of safety: measurement of creatinine | Measured through Month 8
Number of participants with early discontinuation of vaccinations and reason for discontinuation | Measured through Month 8

SECONDARY OUTCOMES:
Response rate of CD4 T-cell responses 2 weeks after the last DNA vaccination | Measured through Month 2.5
  Measured by intracellular cytokine staining (ICS) to the Center for HIV/AIDS Vaccine Immunology (CHAVI) and PTEg peptide pools
Total magnitude of CD4 T-cell responses 2 weeks after the last DNA vaccination | Measured through Month 2.5
  Measured by ICS to CHAVI and PTEg peptide pools
Response rate of CD8 T-cell responses 2 weeks after the last DNA vaccination | Measured through Month 2.5
  Measured by ICS to CHAVI and PTEg peptide pools
Total magnitude of CD8 T-cell responses 2 weeks after the last DNA vaccination | Measured through Month 2.5
  Measured by ICS to CHAVI and PTEg peptide pools
Breadth of CD4 T-cell responses determined by epitope mapping, 2 weeks after the last DNA vaccination | Measured through Month 2.5
  Breadth determined as the number of reactive epitopes to the CHAVI and PTEg peptide pools
Breadth of CD8 T-cell responses determined by epitope mapping, 2 weeks after the last DNA vaccination | Measured through Month 2.5
  Breadth determined as the number of reactive epitopes to the CHAVI and PTEg peptide pools
Response rate of CD4 T-cell responses 2 weeks after each MVA vaccination | Measured through Month 8.5
  Measured by ICS to CHAVI and PTEg peptide pools
Total magnitude of CD4 T-cell responses 2 weeks after each MVA vaccination | Measured through Month 8.5
  Measured by ICS to CHAVI and PTEg peptide pools
Response rate of CD8 T-cell responses 2 weeks after each MVA vaccination | Measured through Month 8.5
  Measured by ICS to CHAVI and PTEg peptide pools
Total magnitude of CD8 T-cell responses 2 weeks after each MVA vaccination | Measured through Month 8.5
  Measured by ICS to CHAVI and PTEg peptide pools
Breadth of CD4 T-cell responses determined by epitope mapping, 2 weeks after MVA vaccination | Measured through Month 8.5
  Breadth determined as the number of reactive epitopes to the CHAVI peptide pools and to PTEg peptide pools
Breadth of CD8 T-cell responses determined by epitope mapping, 2 weeks after MVA vaccination | Measured through Month 8.5
  Breadth determined as the number of reactive epitopes to the CHAVI peptide pools and to PTEg peptide pools
Magnitude of HIV-specific binding immunoglobulin G (IgG) Env antibody (Ab) responses 2 weeks after the last MVA vaccination | Measured through Month 8.5
  Determined by binding Ab multiplex assay (BAMA) and, for a subset, peptide array
Breadth of HIV-specific binding IgG Env Ab responses 2 weeks after the last MVA vaccination | Measured through Month 8.5
  Determined by BAMA and, for a subset, peptide array
Magnitude of HIV-specific binding immunoglobulin A (IgA) Env Ab responses 2 weeks after the last MVA vaccination | Measured through Month 8.5
  Determined by BAMA and, for a subset, peptide array
Breadth of HIV-specific binding IgA Env Ab responses 2 weeks after the last MVA vaccination | Measured through Month 8.5
  Determined by BAMA and, for a subset, peptide array
Magnitude of serum neutralizing antibodies (nAbs) to a panel of standardized HIV-1 isolates | Measured through Month 14
Breadth of serum nAbs to a panel of standardized HIV-1 isolates | Measured through Month 14

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, Study Chair — Brigham and Women's Hospital
Locations (7):
- United States (6):
  - Alabama CRS, Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - Seattle Vaccine and Prevention CRS, Seattle, Washington
- Lausanne Vaccine and Immunotherapy Center CRS, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Moodie Z, Li SS, Giorgi EE, Williams LD, Dintwe O, Carpp LN, Chen S, Seaton KE, Sawant SS, Zhang L, Heptinstall J, Liu S, Grunenberg N, Tomaka F, Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Ake JA, Vasan S, Pantaleo G, Frank I, Baden LR, Goepfert PA, Keefer M, Chirenje M, Hosseinipour MC, Mngadi K, Laher F, Garrett N, Bekker LG, De Rosa S, Andersen-Nissen E, Kublin JG, Lu S, Gilbert PB, Gray GE, Corey L, McElrath MJ, Tomaras GD. A polyvalent DNA prime with matched polyvalent protein/GLA-SE boost regimen elicited the most robust and broad IgG and IgG3 V1V2 binding antibody and CD4+ T cell responses among 13 HIV vaccine trials. Emerg Microbes Infect. 2025 Dec;14(1):2485317. doi: 10.1080/22221751.2025.2485317. Epub 2025 Apr 7. PMID 40190112
- [Derived] Cohen KW, Fiore-Gartland A, Walsh SR, Yusim K, Frahm N, Elizaga ML, Maenza J, Scott H, Mayer KH, Goepfert PA, Edupuganti S, Pantaleo G, Hutter J, Morris DE, De Rosa SC, Geraghty DE, Robb ML, Michael NL, Fischer W, Giorgi EE, Malhi H, Pensiero MN, Ferrari G, Tomaras GD, Montefiori DC, Gilbert PB, McElrath MJ, Haynes BF, Korber BT, Baden LR; NIAID HVTN 106 Study Group. Trivalent mosaic or consensus HIV immunogens prime humoral and broader cellular immune responses in adults. J Clin Invest. 2023 Feb 15;133(4):e163338. doi: 10.1172/JCI163338. PMID 36787249
- [Derived] Campion SL, Brenna E, Thomson E, Fischer W, Ladell K, McLaren JE, Price DA, Frahm N, McElrath JM, Cohen KW, Maenza JR, Walsh SR, Baden LR, Haynes BF, Korber B, Borrow P, McMichael AJ. Preexisting memory CD4+ T cells contribute to the primary response in an HIV-1 vaccine trial. J Clin Invest. 2021 Dec 1;131(23):e150823. doi: 10.1172/JCI150823. PMID 34850742